CLINICAL TRIAL: NCT02645175
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Safety Profile and Ability of TW1025 to Decrease Fatigue
Brief Title: Evaluate the Safety Profile and Ability of TW1025 Oral Solution to Decrease Fatigue
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Meriyana Bio Inc. (Industry)
Collaborators: US Oncology Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TW1025-2014; 13145 (Other: US Oncology Research LLC)
Record Dates: First submitted 2015-12-22; First posted 2016-01-01 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Breast Cancer; Fatigue
Keywords: Paclitaxel; docetaxel; vinorelbine; eribulin
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TW1025 (Experimental): TW1025 oral solution, 20ml, 3 times per day (daily dose: 60 ml)
  Interventions: Dietary Supplement: TW1025
- Placebo (Placebo Comparator): TW1025 oral solution matched placebo, 20ml, 3 times per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: TW1025 — 20ml, 3 times per day (daily dose: 60 ml)
  Other Names: Linease oral solution
  Arms: TW1025
Dietary Supplement: Placebo — 20ml, 3 times per day (daily dose: 60 ml)
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel study to evaluate the safety profile and ability of TW1025 oral solution to decrease fatigue in HER2-negative metastatic breast cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
The study population designed to be enrolled is patients with histologically and/or cytologically confirmed breast cancer with clinical evidence of recurrent or progressive HER2-negative metastatic disease and planning to begin a chemotherapy regimen of physician's choice for HER2-negative MBC who have evidence of fatigue.

An add-on study design to assess the superiority of TW1025 over placebo will be utilized in this study to evaluate whether TW1025 can decrease fatigue in patients with fatigue. The study will be conducted as a double-blind, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* A patient is eligible for the study if all of the following apply:

  1. Female patients at least 18 years of age for study sites in the United States and 20 to 80 years old (inclusive) for study sites in Taiwan
  2. Histologically and/or cytologically confirmed HER2-negative breast cancer with clinical evidence of recurrent or progressive metastatic disease
  3. Patients may have measurable or nonmeasurable metastatic breast cancer.
  4. Planning to begin a new chemotherapy regimen of the physician's choice
  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2
  6. HER2-negative disease per College of American Pathologists (CAP) guidelines (immunohistochemistry (IHC) 0, 1+, or if 2+ fluorescence in-situ hybridization (FISH)-negative ratio < 2.0)
  7. Known ER status: ER-negative (0% of cells positive for ER) or ER-positive (≥1% cells positive for ER) by IHC
  8. Adequate bone marrow function (absolute neutrophil count ≥ 1,500 /µL, hemoglobin count ≥ 8 g/dL, and platelet count > 100,000/µL), total serum bilirubin < 1.5 mg/dL and SGOT/SGPT less than 5-times the upper limit of normal if liver metastases are present or < 2.5-times the upper limit of normal if no liver metastases, and serum creatinine < 1.5 mg/dL
  9. Fatigue score of ≥5 on a 1-to-10 linear analog scale
  10. Pain score of ≤4 on a 1-to-10 linear analog scale
  11. Insomnia score of ≤4 on a 1-to-10 linear analog scale
  12. If of childbearing potential, agrees to use reliable contraceptive method(s) during participation in the study
  13. Estimated life expectancy of at least 6 months
  14. Has provided written informed consent and HIPAA authorization

Exclusion Criteria:

* Any patient meeting any of the exclusion criteria will be excluded from study participation:

  1. Has received radiotherapy or cytotoxic therapy within 3 weeks
  2. Any uncontrolled infection
  3. History of lupus erythematosus, rheumatoid arthritis, ankylosing spondylosis, scleroderma, or multiple sclerosis
  4. History of known brain metastases; Screening for brain metastases is not required
  5. More than 4 prior cytotoxic chemotherapy regimens for metastatic disease
  6. Requirement for ongoing systemic steroid therapy
  7. Currently using any other pharmacologic agents or nonpharmacologic interventions to specifically treat fatigue including psychostimulants, antidepressants, acupuncture, etc.

     Note: Antidepressants used to treat items other than fatigue (such as depression or hot flashes) are allowed if the patient has been on a stable dose for ≥ 3 months and plans to continue for ≥ 1 month. Erythropoietin agents to treat anemia are allowed. Exercise is allowed.
  8. Pain requiring long-acting continuous release narcotic pain medication; however, short-acting opioids (oxycodone, hydrocodone), tramadol, and over the counter analgesics such as acetaminophen or NSAIDs are allowed
  9. Use of any over the counter herbal/dietary supplement marketed for fatigue or energy (for example, products containing any type of ginseng, rhodiola rosea, high doses of caffeine, guarana, or anything called an "adaptogen")
  10. Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily oral TW1025/placebo treatment
  11. Uncontrolled thyroid disorder
  12. Psychiatric disorder such as severe depression, manic depressive disorder, obsessive compulsive disorder or schizophrenia (Defined per medical history)
  13. Any other serious diseases/medical history that would limit the patient's ability to receive study therapy as assessed by the investigator
  14. Lactating, pregnant, or plans to be become pregnant
  15. Has received an investigational agent within 4 weeks of entering this study
  16. History of adverse reactions to any of the ingredients in TW1025.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue scores at 9 weeks post-supplement initiation (+/- 1 week) compared with baseline | Baseline vs 9 weeks
  Change in fatigue scores at 9 weeks post-initiation of supplementation with TW1025/Placebo compared with baseline, assessed by using the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue subscale

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | 1 year after discontinuation of study treatment
  Adverse events (side effects) in each arm will be counted and compared

OTHER OUTCOMES:
Change in Fatigue Scores at Baseline vs at 18-weeks | Baseline vs 18-weeks
  Change in fatigue scores at 18 weeks post-supplement initiation and other on-treatment time points compared with baseline assessed by using the FACIT Fatigue subscale
Change in Sleepiness Scores | Baseline vs 9 weeks
  Change in Daytime sleepiness scores, assessed using the Epworth Sleepiness Scale (ESS)
Change in Quality of Life Scores | Baseline vs 9 weeks
  Change in Quality of life scores, assessed using the Quality of Life Linear Analog Scale (QOL-LAS)
Change in Overall Impression | 9 weeks
  The Subject Global Impression of Change is a 7-point instrument in which the patient rates the change in their overall status since beginning the study drug (ranging from very much better, moderately better, a little better, about the same, a little worse, moderately worse, to very much worse). It has been used extensively for determination of minimally clinically significant differences in numerous oncology clinical trials. Patients will be asked to fill out the Global Impression of Change scale at week 9 after starting study therapy only.
Levels of C-reactive protein in blood | baseline vs 9-weeks vs 18-weeks
  C-reactive protein levels will be measured at baseline, and at weeks 9 and 18 following initiation of dietary supplement.
Change in Gene Expression | Baseline vs 9-weeks vs 18-weeks
  Change in Whole blood gene expression profiles will be assessed using the NanoString® human immunology and the human inflammation gene panels at baseline and at weeks 9 and 18 of dietary supplementation. RNA-Seq or other methodologies may also be utilized to evaluate cytokine and immune cell signaling pathways

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Study Chair — Texas Oncology-Baylor Charles A. Sammons Cancer Center; Jacqueline Whang-Peng, MD., Study Director — Director, Division of Cancer Center, Wan Fang Hospital, Taiwan; Anderson Thomas, MD, Principal Investigator — Texas Oncology-Bedford; Danso Michael, MD, Principal Investigator — Virginia Oncology Associates; Encarnacion Carlos, MD, Principal Investigator — Texas Oncology-Waco; Fleischauer Scott, MD, Principal Investigator — Texas Oncology-Arlington North; Taguchi Julie, MD, Principal Investigator — Sansum Clinic; Wang Grace, MD, Principal Investigator — Baptist Health Medical Group Oncology, LLC; Holmes Frankie, MD, Principal Investigator — Texas Oncology-Memorial City; Houck William, MD, Principal Investigator — Shenandoah Oncology, P.C.; Crane Gregory, MD, Principal Investigator — The University of Kansas Cancer Center; Tsai Michaela, MD, Principal Investigator — Minnesota Oncology Hematology, P.A.; Vukelja Svetislava, MD, Principal Investigator — Texas Oncology-Tyler; Lee Jae, MD, Principal Investigator — Willamette Valley Cancer Institute and Research Center; Smith II John, MD, Principal Investigator — Northwest Cancer Specialists, P.C.

IPD SHARING:
Plan to Share IPD: Yes
Each study site has at least three monitors for the study and all of data will send to Data Center in DSG immediately for all study physicians reference.

REFERENCES:
- See also: Evaluation of the Safety and Efficacy of THL-P in Metastatic Breast Cancer — https://clinicaltrials.gov/ct2/show/NCT00976365